CLINICAL TRIAL: NCT06228352
Title: Is Clostridioides Difficile Infection Associated With Changes in Bile Acid Profiles in Children With Ulcerative Colitis
Brief Title: Role of Bile Acids and Microbiota in Clostridioides Difficile Infection in Ulcerative Colitis
Acronym: ABRICO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221179; 2022-A01579-34 (Other: IDRCB Number)
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Clostridioides difficile infection; Intestinal dysbiosis; Bile acid profiles
MeSH Terms: conditions — Colitis, Ulcerative; Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ulcerative colitis flare-up: Patient with ulcerative colitis, whatever the extent, except isolated proctitis (<5 cm), diagnosed for more than 3 months, presenting with a flare of UC defined by a Pediatric Ulcerative Colitis Activity Index (PUCAI) score between 35 and 65.
  Interventions: Other: Feces collection
- Ulcerative colitis remission: Patient with ulcerative colitis, whatever the extent, except isolated proctitis (<5 cm), diagnosed for more than 3 months and in clinical remission defined by a Pediatric Ulcerative Colitis Activity Index (PUCAI) score under 10.
  Interventions: Other: Feces collection
- Controls: Paediatric patients (<18 years) without chronic liver disease or chronic digestive disease (celiac disease, inflammatory bowel disease, chronic diarrhea) and hospitalized for an endoscopic examination to investigate abdominal pain, gastroesophageal reflux or polyposis.
  Interventions: Other: Feces collection

INTERVENTIONS:
Other: Feces collection — A single stool sample will be taken (a specific kit will be given to the patient for this) during a consultation for follow-up or hospitalization.
  Stool samples will be used to study the composition of the intestinal microbiota and to measure faecal biomarkers.

SUMMARY:
Ulcerative Colitis (UC) is a chronic Inflammatory Bowel Disease characterized by chronic inflammation of the colon. Composition of gut microbiota of UC patients is abnormal (dysbiosis).

Ulcerative Colitis patients have an increased risk of Clostridioides difficile infection (CDI) and CDI complications (colectomy, death, recurrence). The reason for this increased risk in IBD patients is not fully understood. The decrease in the proportion of secondary bile acids, induced by microbiota dysbiosis in patients with UC could favor C. difficile infection.

The main objective of the study is to describe the composition of bile acids (primary and secondary) in children followed for UC during relapse with or without CDI and to compare it to children with UC in remission and healthy controls. The composition of fecal microbiota will be also describe to correlate dysbiosis and bile acid abnormalities. And finally some fecal biomarkers will be study : short chain fatty acids, metabolic pathway of Tryptophan, and fecal Calprotectin.

DETAILED DESCRIPTION:
Ulcerative Colitis (UC) is a chronic inflammatory bowel disease (IBD) characterized by chronic inflammation of the colon. Clinical symptoms include bloody diarrhea associated with abdominal pain, fecal incontinence, urgency, and tenesmus. Approximately 15-20% of patients develop UC during childhood or adolescence, with a sustained worldwide rise of the incidence of IBD, particularly pediatric forms. While there are many similarities between adult- and childhood-onset UC, pediatric-onset UC appears to be more severe and extensive with more rapid spread of the disease leading to high morbidity, more severe acute flares and more frequent use of intravenous corticosteroids. To date, there is no medical treatment that can cure the disease but only treatments that shorten the duration of relapses or prevent them.

An imbalance in the composition of the intestinal microbiota named "dysbiosis" has been demonstrated in IBD. This dysbiosis is characterized by a strong instability of the microbiota over time, and a reduction of diversity and particularly a reduction in bacteria belonging to the Firmicutes and Bacteroidetes phyla with an increase in Proteobacteria and Actinobacteria. More recently, a UC-specific dysbiosis has been described including a decrease in butyrate-producing bacteria, in particular Faecalibacterium prausnitzii, and Roseburia hominis.

It has also been shown that if adult patients with UC in flare-up and remission have similar total fecal bile acids, they have a lower proportion of fecal secondary acids compared to healthy control subjects.

Patients with UC have an increased risk of Clostridioides difficile infection (CDI) and complications from the CDI (coletomy, deaths) as well as a higher risk of CDI recurrences. Clostridioides difficile is a strict anaerobic bacteria, which represents the main cause of post-antibiotic diarrhea.

The hypothesis of the project is that gut microbiota dysbiosis in patients with UC alters the bile acid profile and metabolite profile and could promote C difficile infection in these patients without any other risk factors such as antibiotics. To confirm this hypothesis, the investigating team proposes to study the microbiota, bile acid profiles and microbial metabolites in the stools of 40 pediatric-onset UC patients with a flare-up of their disease with (n=20) or without (n=20) a concomitant CDI and to compare them to healthy children (n=20) and UC children with clinical remission (n=20). Bile acids will be determined by high performance liquid chromatography coupled with tandem mass spectrometry detection, the short chain fatty acids and tryptophan derivatives derived from TRP and AGCC will be determined by GC-MS or LC-MS and the microbiota by the MiSeq technique.

The investigating team hopes to identify bile acid profiles predisposing for CDI and to correlate them with microbiota abnormalities. This will allow to better understand the factors associated with CDI but also to identify biomarkers of infection and maybe protective bacterial strains. In the long term, the investigating team hopes to find new therapeutic perspectives by providing bacteria of interest to transform bile acids and to protect against Clostridioides difficile.

ELIGIBILITY:
For everyone :

Inclusion Criteria:

* Pediatric patients (<18 years) consultant or hospitalized in the Gastroenterology department of Necker-Enfants Malades Hospital.
* Information and consent of parents and the patient

Exclusion Criteria:

* Patient who received antibiotic or antifungal treatment in the 4 weeks prior to inclusion.
* Patients colonized by C. difficile.
* Pregnant or breastfeeding young girl.
* Refusal of the protocol by parents or patient.

For group 1: Patients with active UC

Inclusion criteria:

* Patient with UC, whatever the extent, except isolated proctitis (<5 cm), diagnosed for more than 3 months according to the usual clinical, biological and endoscopic criteria.
* UC in flare defined by a PUCAI score of between 35 and 65.

Non-inclusion criteria:

* Patient with IBD unclassified or Crohn's disease.
* Patient with isolated proctitis (<5 cm).
* Colectomized patients.
* Patients with sclerosing cholangitis associated with their UC or liver disease.

Group 2: Patients in UC remission

Inclusion criteria:

* Patient with UC, whatever the extent, except isolated proctitis (<5 cm), diagnosed for more than 3 months according to the usual clinical, biological and endoscopic criteria.
* UC in remission defined by a PUCAI score <10.

Non-inclusion criteria:

* Patient with IBD unclassified or Crohn's disease.
* Patient with isolated proctitis (<5 cm).
* Colectomized patients.
* Patients with sclerosing cholangitis associated with their UC or liver disease.

Group 3: Healthy control subjects

Inclusion criteria:

- Patients hospitalized for an endoscopic assessment to control for abdominal pain, gastroesophageal reflux or polyposis.

Non-inclusion criteria:

* Patient with chronic liver disease.
* Patient with chronic digestive disease (celiac disease, IBD, chronic chronic).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients consulting or hospitalized in the Gastroenterology department of Necker-Enfants Malades Hospital, with ulcerative colitis (UC) in flare-up with and without Clostridioides difficile infection (CDI), patients UC in remission and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composition of bile acids | Day 0
  Description of the composition of primary and secondary bile acids. Fecal bile acids will be assayed by high performance liquid chromatography coupled with detection by tandem mass spectrometry and the quantification of each bile acid will be expressed as a percentage of total bile acids.
  The bile acid profile of the patients will be compared between the 3 groups: patients followed for ulcerative colitis (UC) in flare with or without a concomitant C difficile infection, patients with UC in clinical remission and healthy subjects without UC.

SECONDARY OUTCOMES:
Faecal microbiota | Day 0
  The composition of the patients' faecal microbiota will be measured by targeted metagenomics (high-throughput sequencing of DNA coding for 16S RNA targeting the V3-V4 region). The analysis of the diversity of the microbiota will be carried out by calculating the Shannon index. This index will be compared between the groups with and without CDI.
Short-chain fatty acids | Day 0
  Analysis of fecal biomarkers. Short-chain fatty acids (SCFAs; acetate, propionate, butyrate and branched short-chain fatty acids) and metabolites of the tryptophan pathway will be determined by gas or liquid chromatography methods, coupled with mass spectrometric detection. The results will be compared between the 3 groups.
Metabolic pathway of tryptophan | Day 0
  Analysis of fecal biomarkers. Metabolites of tryptophan pathway will be determined by gas or liquid chromatography methods, coupled with mass spectrometric detection The results will be compared between the 3 groups.
Fecal calprotectin | Day 0
  Analysis of fecal biomarkers. Fecal calprotectin assay will be done by chemiluminescence assay. The results will be compared between the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte Pigneur, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Frédéric Barbut, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No